CLINICAL TRIAL: NCT02729701
Title: Pilot Study of the Effect of Duavee® on Benign Breast Tissue Proliferation in Peri or Post-menopausal Women at Moderate Risk for Development of Breast Cancer
Brief Title: Pilot Study of the Effect of Duavee® on Benign Breast Tissue Proliferation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Center, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002440
Record Dates: First submitted 2016-03-21; First posted 2016-04-06 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estrogens, Conjugated (USP); bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duavee (Experimental): Participants will be asked to take Duavee for 6 months while on the study.
  Interventions: Drug: Duavee

INTERVENTIONS:
Drug: Duavee — Once daily tablet of Duavee (Bazedoxifene (20 mg) plus conjugated estrogen (0.45 mg))
  Other Names: conjugated estrogens/bazedoxifene

SUMMARY:
The purpose of this study is to learn whether daily use of Duavee® is accepted and tolerated by peri- and post-menopausal women at moderate risk for development of breast cancer.

DETAILED DESCRIPTION:
Duavee® is tissue specific estrogen complex of bazedoxifene plus conjugated estrogen which is FDA approved for relief of menopausal symptoms and prevention of osteoporosis in women with a uterus who have not been diagnosed with estrogen dependent neoplasia. The overall purpose of this research is to demonstrate in a preliminary fashion that despite reduction in menopausal symptoms, (Duavee®) does not increase and may decrease proliferation in benign breast tissue in a cohort of peri- or post-menopausal women at moderately increased risk for breast cancer. If this pilot shows rapid accrual, good retention, and lack of significant increase in the risk biomarker Ki-67 in benign breast tissue, a larger prevention trial is envisioned

ELIGIBILITY:
Inclusion Criteria:

* Women with vasomotor symptoms with a uterus who are postmenopausal or in late menopause transition
* Body Mass Index (BMI) <36 kg/m2
* Class I-III mammogram within 6 months of Random Periareolar Fine Needle Aspiration (RPFNA); If Class 0 or 4, must be resolved with additional procedures
* If previously on oral contraceptives or hormone replacement, off for 8 weeks or more prior to baseline RPFNA; the exception is low dose vaginal hormones
* Confirmed moderate risk of developing breast cancer
* RPFNA results within study defined range
* Kidney and liver function within study defined range
* Willing and able to comply with study related procedures

Exclusion Criteria:

* Previous biopsy showing evidence of breast cancer
* Have a predisposition to or prior history of thromboembolism, deep venous thrombosis, pulmonary embolism, or stroke
* History of renal or liver disease
* Prior ovarian or endometrial cancer
* Stopped or started hormone replacement within 8 weeks
* Any other condition or intercurrent illness that in the opinion of the investigator makes the woman a poor candidate for RPFNA
* Currently taking or have taken specific medications in the past 6 months
* Participation on any chemoprevention trial within 6 months
* Current illness which would make potential participant unsuitable for enrollment

Max Age: 61 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center Breast Cancer Prevention Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in aggregate; no individual participant data will be made available.
Supporting Information: Study Protocol
Time Frame: 2021-2022
Access Criteria: upon request.

REFERENCES:
- [Result] Fabian CJ, Nye L, Powers KR, Nydegger JL, Kreutzjans AL, Phillips TA, Metheny T, Winblad O, Zalles CM, Hagan CR, Goodman ML, Gajewski BJ, Koestler DC, Chalise P, Kimler BF. Effect of Bazedoxifene and Conjugated Estrogen (Duavee) on Breast Cancer Risk Biomarkers in High-Risk Women: A Pilot Study. Cancer Prev Res (Phila). 2019 Oct;12(10):711-720. doi: 10.1158/1940-6207.CAPR-19-0315. Epub 2019 Aug 16. PMID 31420361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the Breast Cancer Prevention Center. Accrual May 2016 - August 2018. 42 women were considered medically eligible and were screened by Random Periareolar Fine Needle Aspiration (RPFNA). 14 did not enter the trial for a variety of reasons.
Groups:
- Duavee: Participants asked to take Duavee for 6 months while on the study.
  Duavee: Once daily tablet of Duavee (Bazedoxifene (20 mg) plus conjugated estrogen (0.45 mg))
Period: Overall Study
Arm/Group | Duavee
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Duavee
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 53 [45 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Proliferation Index (percent of breast epithelial cells that are Ki-67 immunocytochemistry positive) [Median (Full Range); unit: percent] | 1 [0 to 3.6]
Fibroglandular Volume (FGV) [Median (Full Range); unit: cm-squared] — total fibroglandular volume for both breasts derived from assessment of mammograms using the Volpara(R) software program.
  cm-squared | 133 [36 to 336]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility for a Larger Trial
Description: Outcome will be based on three separate factors used collectively to determine feasibility of the study and consideration of a subsequent larger trial. These are accrual rate (ability to accrue target number of subjects in a timely manner), dropout rate (frequency of subjects who are compliant and complete the intervention) and change in Ki-67 (increase vs decrease in percent of cells stained positive in the majority of subjects). Should accrual be inadequate or too slow; or if retention is too low; then a decision would be made not to proceed to a larger trial. Also, if there is evidence of an increase in proliferation (Ki-67) then no further studies would be planned.
Time Frame: 6 Months
Population: potential subjects screened for eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavee
Number analyzed (Participants) | 42
Participants
  Screened | 42
  Eligible | 28
  Complete | 28

2. Secondary Outcome: Change in Ki-67
Description: Assessment by immunocytochemistry of the percent of breast epithelial cells staining positive.
  Per protocol, restricted to those subjects with baseline Ki-67 positivity >1.0% but < 4%
Time Frame: Change from Baseline to Month 6
Population: All subjects with baseline Ki-67 >1%
Measure: Median (Full Range); unit: change in percent positivity
Arm/Group | Duavee
Number analyzed (Participants) | 15
change in percent positivity | -1.2 [-3.2 to 3.2]
Statistical Analysis 1: Comparison: Duavee; Test for within-group change by paired two-sample non-parametric test; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance <0.05

3. Secondary Outcome: Change in Fibroglandular Volume (FGV)
Description: Assessment of mammograms for percent of breast defined as FGV by Volpara automated assessment.
Time Frame: Change from Baseline to Month 6
Population: Subjects with baseline and post-intervention mammograms assessed by Volpara
Measure: Median (Full Range); unit: cm-squared
Arm/Group | Duavee
Number analyzed (Participants) | 26
cm-squared | -12 [-204 to 62]
Statistical Analysis 1: Comparison: Duavee; Test for within-group change via paired, two-sample non-parametric test; Test type: Other; p = 0.043, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance <0.05; 2-sided

4. Secondary Outcome: Change in Body Composition (Total Mass)
Description: Assessment by Dual Energy X-ray Absorptivity (DEXA)
Time Frame: Change from Baseline to Month 6
Population: All subjects enrolled and completed
Measure: Median (Full Range); unit: kg
Arm/Group | Duavee
Number analyzed (Participants) | 28
kg | 0.9 [-11.8 to 10.4]
Statistical Analysis 1: Comparison: Duavee; Test for within-group change using paired two-sample non-parametric etst; Test type: Other; p = 0.088, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance < 0.05

5. Secondary Outcome: Levels of Bazedoxifene in the Blood
Description: Assessment of concentration of bazedoxifene in plasma by High-performance liquid chromatography (HPLC)
Time Frame: Month 6
Population: With residual plasma available for analysis
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Duavee
Number analyzed (Participants) | 25
ng/ml | 1.83 [0.004 to 7.86]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Self-reported adverse events
Arm/Group | Duavee
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
Pfizer, Inc. provided the study agent Duavee but was otherwise not involved in the design, conduct, or analysis of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02729701/Prot_SAP_000.pdf